CLINICAL TRIAL: NCT01321866
Title: Randomized Trial Comparing a Cutting Balloon to a Non-cutting Balloon for the Treatment of Venous Stenosis in the Fistulas of Hemodialyzed Patients
Brief Title: Cutting Balloon Versus Non-cutting Balloon for the Treatment of Venous Stenosis in the Fistulas of Hemodialyzed Patients
Acronym: PREST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion curve too slow.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AOI/2010/EP-01; 2011-A00332-39 (Other: RCB number)
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Arteriovenous Fistula; Fistula
Keywords: Angioplasty; cutting balloon
MeSH Terms: conditions — Arteriovenous Fistula; Fistula | interventions — Angioplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental arm (Experimental): Patients in this arm will have angioplasty of a fistula stenosis using a cutting balloon
  Interventions: Procedure: Cutting balloon angioplasty
- Standard arm (Active Comparator): Patients in this arm will have angioplasty of a fistula stenosis using a non-cutting balloon.
  Interventions: Procedure: Angioplasty

INTERVENTIONS:
Procedure: Cutting balloon angioplasty — Angioplasty of fistula stenosis using a cutting balloon
  Arms: Experimental arm
Procedure: Angioplasty — Angioplasty of fistula stenosis using a non-cutting balloon
  Arms: Standard arm

SUMMARY:
The main objective of this study is to evaluate and compare the primary patency rate at 12 months in a group of hemodialysis patients operated on by cutting balloon and in a group of hemodialysis patients operated by conventional balloon.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 12 months of follow-up
* The patient is on hemodialysis because of chronic renal insufficiency
* The patient's vascular access is an arterio-venous fistula
* The patient has a venous stenosis in the fistula (first event in the studied zone)
* The patient is scheduled for angioplasty

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient cannot fluently read French
* The patient cannot understand French
* The patient is pregnant
* The patient is breastfeeding
* Short term dialysis
* The vascular access is a "graft"
* The stenosis in question is a recurrence, and not a first event in the studied zone
* The life expectancy of the patient is < 12 months
* Medical emergency situation
* Peritoneal dialysis
* At-home dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Primary patency | 12 months
  Primary patency following a first angioplasty of a first stenose in the affected zone.

SECONDARY OUTCOMES:
Number of early re-stenoses | 3 months
  stenosis defined as lumen diameter < 2mm
Number of re-stenoses | 12 months
  Stenosis defined as lumen diameter < 2mm
Total days in hospital | 12 months
  The total number of days hospitalized for stenosis, thrombosis, or recovering vascular access. This does not include regular hemodialysis activities.
Number of stents used | 12 months
  The total number of stents placed between the study angioplasty and the end-of-study visit.
Total number of venous thromboses | 12 months
  Total number of venous thromboses between study angioplasty and end-of-study visit
Direct medical costs (€) | 12 months
Indirect costs (€) | 12 months
Questionnaire KDQOL | 12 months
Questionnaire SF36 | 12 months
Questionnaire KDQOL | 3 months
Questionnaire KDQOL | 6 months
Questionnaire SF36 | 3 months
Questionnaire SF36 | 6 months
Fistula quality (cm*ml/min) | Baseline
  cumulative length of "usable" fistula (cm) * venous flow during the last hemodialysis (ml/min)
Fistula quality (cm*ml/min) | 6 months
  cumulative length of "usable" fistula (cm) * venous flow during the last hemodialysis (ml/min)
Fistula quality (cm*ml/min) | 12 months
  cumulative length of "usable" fistula (cm) * venous flow during the last hemodialysis (ml/min)
% Stenosis | Baseline
  100-((the smallest diameter of the stenosis lumen (mm)/ the diameter of a proximal, normal portion of lumen (mm))*100)
% Stenosis | 6 months
  100-((the smallest diameter of the stenosis lumen (mm)/ the diameter of a proximal, normal portion of lumen (mm))*100)
% Stenosis | 12 months
  100-((the smallest diameter of the stenosis lumen (mm)/ the diameter of a proximal, normal portion of lumen (mm))*100)
Presence/absence of complications associated with the angioplasty | Day of intervention
% Stenosis | 3 months
  100-((the smallest diameter of the stenosis lumen (mm)/ the diameter of a proximal, normal portion of lumen (mm))*100)
Presence/absence of complications since the last visit | 6 months
Presence/absence of complications since the last visit | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Picard, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France